CLINICAL TRIAL: NCT01250483
Title: Effects of Alpha Blockers on Prostate-specific Antigen (PSA) Change in Men With Lower Urinary Tract Symptoms (LUTS)
Status: Completed | Type: Observational
Sponsor: Seoul National University Hospital (Other)
Other Study IDs: PSA and alpha blockers
Record Dates: First submitted 2010-11-25; First posted 2010-11-30 (Estimated); Last update posted 2010-11-30 (Estimated); Status verified 2010-11

CONDITIONS: Benign Prostatic Hyperplasia; Prostate Cancer
Keywords: prostate; prostate-specific antigen; benign prostatic hyperplasia; adrenergic alpha-Antagonists
MeSH Terms: conditions — Prostatic Hyperplasia; Prostatic Neoplasms | interventions — Prostate-Specific Antigen

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- BPH: men aged more than 40 years who presented with BPH/LUTS and showed negative results of transrectal prostate biopsy before the period of AB medication
  Interventions: Other: PSA measurement, uroflowmetry, IPSS, transrectal ultrasonography
- prostate cancer: men aged more than 40 years who presented with BPH/LUTS and showed positive results of transrectal prostate biopsy before the period of AB medication
  Interventions: Other: PSA measurement, uroflowmetry, IPSS, transrectal ultrasonography

INTERVENTIONS:
Other: PSA measurement, uroflowmetry, IPSS, transrectal ultrasonography

SUMMARY:
The correlation between the change of serum prostate-specific antigen (PSA) or PSA velocity (PSAV) and severity of lower urinary tract symptoms (LUTS) has been poorly understood. Previous studies usually focused on the treatment efficacy or preventive role of alpha blockers (AB) for clinical progression of benign prostatic hyperplasia (BPH) and AB therapy in real-life practice improved BPH/LUTS and reduced the risk of overall clinical progression. We hypothesized that the change of PSA and PSA velocity would be correlated to LUTS severity in the groups of BPH and prostate cancer.

DETAILED DESCRIPTION:
Since successful treatment with alpha-1 adrenergic antagonists, or AB was reported first in 1975, the therapeutic efficacy has been widely accepted and now AB medication is considered the first-line choice worldwide among pharmacologic options for BPH-related LUTS.

Previous studies usually focused on the treatment efficacy or preventive role of AB for clinical progression of BPH and AB therapy in real-life practice improved BPH/LUTS and reduced the risk of overall clinical progression. However, the correlation between the change of serum PSA or PSAV and severity of LUTS has been poorly understood. Some studies showed follow-up data of PSA during the study period, and they failed to show a significant change of PSA in the group of AB. In contrast, some other studies demonstrated that the possibility of PSA change with the presence of LUTS and it is early to tell conclusively that there would be no relationship between PSA values and LUTS severity. Because a PSA value is considered an important factor to determine whether transrectal prostate biopsy should be performed, We hypothesized that the change of PSA and PSAV would be correlated to LUTS severity in the groups of BPH and prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* more than two consecutive PSA measurements before the biopsy and the medication periods of AB more than 3 months in all patients

Exclusion Criteria:

* any prostate surgery during the study period, any prostate disease with evidence of prostatic inflammation, any urologic surgery before PSA measurement, and medication history of anticholinergics or 5-alpha reductase inhibitors

Ages: 40 Years to 80 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Men aged more than 40 years who presented with BPH/LUTS and performed transrectal prostate biopsy during the period of AB medication between January 2001 and December 2009.
Sampling Method: Probability Sample
Enrollment: 174 (Actual)
Dates: Start 2001-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
PSAV | calculated PSAV using baseline PSA value and PSA 6 month or 1 year after initial PSA measurement
  PSAV values were calculated by a simple method: [(last PSA values - initial PSA values)/measurement period (month)]

SECONDARY OUTCOMES:
international prostate symptoms symptom score (IPSS), maximal flow rate (Qmax) | IPSS scores and Qmax values at the time of baseline PSA measurement and 6 month or 1 year after initial PSA measurement
  IPSS scores, quality of life (QOL) scores of IPSS questionnaire (Question 8), and maximal flow rates (Qmax)

CONTACTS AND LOCATIONS:
Overall Officials: Cheol Kwak, M.D.,Ph.D., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea